CLINICAL TRIAL: NCT03929380
Title: Acute Effects of Squat Protocols in Muscular Power, Postural Sway and Tendinous Thickness.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid situation
Sponsor: Iñigo Fernández de Luco Santamaría (Other)
Responsible Party: Sponsor-Investigator, Iñigo Fernández de Luco Santamaría, Doctoral Student, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 662550
Record Dates: First submitted 2019-04-22; First posted 2019-04-26 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Acute Squat Training Effects
Keywords: Squat; Acute effect; Tendon thickness; Counter movement jump test; Postural sway; Muscular power

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10x10 squat protocol (Experimental)
  Interventions: Other: Squat protocol
- As Fast As Possible 100 squat protocol (Experimental)
  Interventions: Other: Squat protocol

INTERVENTIONS:
Other: Squat protocol — 60% of 1RM weight for 100 squat reps

SUMMARY:
The objective of this study is to know the acute effects of a squat protocol in: 1- lower limb muscle power analyzed by countermovement jump on force platform and upper limb through a bench press with encoder test; 2 - the unipodal postural equilibrium by force platform; 3 - the patellar tendinous thickness measured by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Males, with at least a year of experience in heavylift exercises, age between 20 and 35 years.

Exclusion Criteria:

-

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 0 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Muscle power | 30 minutes
  Muscle power of lower limbs measured by countermovement jump on force platform
Patellar thickness | 60 minutes
  Tendon thickness of the patellar tendon measured by ultrasound
Monopodal Postural Sway | 10 minutes
  Monopodal postural balance with open eyes in force platform

SECONDARY OUTCOMES:
Muscular fatigue | 30 minutes
  Muscle fatigue measured in each resting period by means of a countermoving jump to assess the loss of power.

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier Orquín Castrillón, Study Director — Universidad Católica San Antonio de Murcia; Iñigo Fernández de Luco Santamaría, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- UCAM Sports Center, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Butcher S. J, Judd T. B, Benko C. R, Horvey K. J, Pshyk A. D, (2015). Relative intensity of two types of crossfit exercise: Acute circuit and high-intensity interval exercise. Journal of Fitness Research, 4 (2), 3-15.
- [Background] Fredberg U, Bolvig L, Andersen NT, Stengaard-Pedersen K. Ultrasonography in evaluation of Achilles and patella tendon thickness. Ultraschall Med. 2008 Feb;29(1):60-5. doi: 10.1055/s-2007-963027. Epub 2007 Aug 16. PMID 17703377
- [Result] Fisker FY, Kildegaard S, Thygesen M, Grosen K, Pfeiffer-Jensen M. Acute tendon changes in intense CrossFit workout: an observational cohort study. Scand J Med Sci Sports. 2017 Nov;27(11):1258-1262. doi: 10.1111/sms.12781. Epub 2016 Oct 7. PMID 27714843
- [Result] Mate-Munoz JL, Lougedo JH, Barba M, Garcia-Fernandez P, Garnacho-Castano MV, Dominguez R. Muscular fatigue in response to different modalities of CrossFit sessions. PLoS One. 2017 Jul 28;12(7):e0181855. doi: 10.1371/journal.pone.0181855. eCollection 2017. PMID 28753624